CLINICAL TRIAL: NCT01381393
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety of BONVIVA(Ibandronate) Administered in Korean Patients According to the Prescribing Information
Brief Title: BONVIVA(Ibandronate) PMS(Post-marketing Surveillance )
Acronym: BONPMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110603
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Osteoporosis
Keywords: osteoporosis; ibandronate
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ibandronate: The subjects with osteoporosis in postmenopausal women
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Basically there is no treatment allocation. Subjects who would be administered of ibandronate at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.
  Other Names: BONVIVA

SUMMARY:
This is an open label, multi-centre, non-interventional post-marketing surveillance.

DETAILED DESCRIPTION:
This is an open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety of ibandronate administered in Korean patients according to the prescribing information.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

1. Subjects diagnosed with osteoporosis in postmenopausal women.
2. Subjects who the investigator believes that they can and will comply with the requirements of the protocol
3. Subjects with no experience of treatment using ibandronate.
4. Subjects who are administered of ibandronate in normal prescription use

Exclusion Criteria:

Considering the nature of this non-interventional PMS study, there is no strict exclusion criteria set up. The doctors participating this study to enrol the subjects prescribed with ibandronate following the locally approved Prescribing Information.

The following criteria should be checked at the time of study entry.

According to contraindication on the prescribing information, ibandronate should not be administered to the following patients:

1. Patients with known hypersensitivity to ibandronate or to any of its excipients
2. Uncorrected hypocalcemia
3. Inability to stand or sit upright for at least 60 minutes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated ibandronate with postmenopausal osteoporosis in Korea
Sampling Method: Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2007-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The number of adverse event after ibandronate administration | 6 months

SECONDARY OUTCOMES:
The number of unexpected adverse events after ibandronate administration | 6 months
The number of serious adverse events after ibandronate administration | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea